CLINICAL TRIAL: NCT04904822
Title: Abdominal Versus Vaginal Uterine Bisection for Retrieval of Large Uteri During Laparoscopic Hysterectomy: A Randomized Controlled Study
Brief Title: Abdominal Versus Vaginal Bisection in Laparoscopic Hysterectomy
Acronym: TLH-Bisection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Ayman S Dawood, MD, Assistant professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: uterine bisection
Record Dates: First submitted 2021-05-24; First posted 2021-05-27 (Actual); Last update posted 2024-03-13 (Actual); Status verified 2024-03

CONDITIONS: Hysterectomy; Laparoscopy; Uterine Bisection; Large Uteri

STUDY DESIGN:
Intervention Model Description: 2 groups parallel allocation
Who Masked: Participant
Masking Description: Closed envelopes containing allocations
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Vaginal bisection of uterus
  Interventions: Procedure: Vaginal bisection
- Control group (Experimental): Abdominal bisection
  Interventions: Procedure: Abdominal bisection

INTERVENTIONS:
Procedure: Vaginal bisection — Uterine bisection vaginally by scalpel 24
  Arms: Study group
Procedure: Abdominal bisection — Uterine bisection by endokinfe
  Arms: Control group

SUMMARY:
Large uteri present a challenge during Total lap.hysterectomy and its extraction is another challenge. This study addressees and compare 2 methods of retrieval of large uteri

DETAILED DESCRIPTION:
Despite a number of publications about TLH for large uterus, few surgeons have compared the results of their technique of TLH through the vagina or abdominal bisection. The aim of this study was to compare the clinical results of TLH for large uterus through transvaginal or abdominal bisection approaches after strict preoperative assessment.

ELIGIBILITY:
Inclusion Criteria:

* large uterus ≥ 12weeks,
* benign pathology,
* mobile uterus
* BMI less than 30kg/m2

Exclusion Criteria:

* unfit for laparoscopy,
* Extensive pelvic adhesions,
* Extensive endometriosis
* malignancy
* virgin cases

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Retrieval time of uterus | 6 months
  Time from end of colpotomy to extraction of uterus
Blood loss | 6 months
  Amount of blood in suction

SECONDARY OUTCOMES:
Injury of other organs | 6 months
  Number of cases with intraoperative injuries

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
we will share results and statistical analysis on valuable request
Supporting Information: Study Protocol, SAP
Time Frame: 3 months